CLINICAL TRIAL: NCT05857189
Title: Assessment of the Quality-of-life Impact of Newly Formed Digitalized Printed Paper Inserted Into Eyeglasses for Unilateral Eye Defect Patient Rehabilitation (Clinical Trial)
Brief Title: Quality-of-life Impact of Newly Formed Digitalized Printed Paper Inserted Into Eyeglasses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: QoL_2022
Record Dates: First submitted 2023-04-02; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Orbital Deformity

STUDY DESIGN:
Intervention Model Description: Crossover between experimental and traditional groups after 2 weeks of lapse time. both groups will be compared to healthy control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental)
  Interventions: Device: Digitalized printed paper
- Control group (Active Comparator)
  Interventions: Device: Traditional drawing image
- Healthy control group (Other): patients in this group will be observed as a normal reference group
  Interventions: Other: Healthy controls

INTERVENTIONS:
Device: Digitalized printed paper — Patients will receive a newly formed digitalized printed paper inserted into eyeglasses
  Arms: Experimental group
Device: Traditional drawing image — Patients will receive eyeglasses that hold a traditional drawing image of the eye
  Arms: Control group
Other: Healthy controls — Patients will include volunteering participants with un defected eye
  Arms: Healthy control group

SUMMARY:
A straightforward, user-friendly removable orbital prosthesis is a practical choice for effective rehabilitation in such patients with defective eyes. One of the essential elements for a good recovery is the retention of the prosthesis. The prosthesis can be retained by using a spectacle frame, conformers, adhesives, osseointegrated implants, magnets, or buttons. Only osseointegrated prostheses in the maxillofacial region can use semi-precision attachments.

DETAILED DESCRIPTION:
Aim: Using of eyeglasses with newly formed digitalized printed paper of mirrored photograph of an intact eye for orbital defected patients to restore the esthetic appearance. An evaluation of the quality of life for patients using temporalized eyeglasses with digitalized printed paper of mirrored photographs of a healthy eye.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an orbital defective eye (type I).
* Patients age more than 6 years.
* Patients with a unilateral enucleated eye.
* Skin-grafted orbital defects with a lack of natural retentive means either natural undercuts or retaining implants.
* Patients who are not prone to be received any prosthetic rehabilitation either for financial, age, or transportation problems of material that are needed for fabrication of prosthetic eye.

Exclusion Criteria:

* Patients with the bilateral enucleated eye.
* Patients with primary signs of skin inflammation, infection, or untreated local disease
* Patients refusing to wear any eyeglasses.
* Patients with ocular defects.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life score | Through study completion, average 6 months
  each person's medical chart. Participants will complete the Arabic version of the World Health Organization Quality of Life Instrument, Short Form (WHOQOL-BREF) before and after intervention.
  The 26- item WHOQOL-BREF Arabic version consists of two overall items measuring general QOL and health condition and 24 items that are universally adopted for the WHOQOL-BREF in four domains: physical health, psychological health, social relationships, and environment. Each item will be rated on a 5- point Likert scale and the domain scores were transformed on a scale from 0 to 100
Patient behaviour toward using the newly designed eye glasses | Through study completion, average 6 months
  The 14-item visual function questionnaire (VF-14), is based on 14 vision-dependent activities performed in everyday life, and the difficulty undertaking each activity is rated Scores range from 0 to 100, and higher scores represent better visual functioning and less difficulty to perform daily activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt